CLINICAL TRIAL: NCT03007654
Title: Evaluate Anti-adhesive Effect and Safety of a Mixed Solid of Poloxamer, Gelatin and Chitosan(Mediclore®) for Intraperitoneal Adhesion in Patient With Gynecological Surgery, a Multicenter Single-blinded, Randomized Study
Brief Title: Evaluate Anti-adhesive Effect and Safety of a Mixed Solid of Poloxamer, Gelatin and Chitosan(Mediclore®)
Acronym: antiadhesion
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yong Sang Song (Other)
Responsible Party: Sponsor-Investigator, Yong Sang Song, MD, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CG-AHS008
Record Dates: First submitted 2016-12-30; First posted 2017-01-02 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Gynecologic Disease
MeSH Terms: conditions — Genital Diseases, Female

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mediclore (Experimental): adhesion barrier Mediclore 5cc, to apply medical device fully around surgery area
  Interventions: Device: Mediclore
- No treatment (No Intervention): standard treatment for surgery
- Adept (Active Comparator): adhesion barrier, Adept, to apply medical device fully around surgery area
  Interventions: Device: Adept

INTERVENTIONS:
Device: Mediclore — apply medical device fully around intrauterine surgery area
  Other Names: Poloxamer, Gelatin and Chitosan.
  Arms: Mediclore
Device: Adept — apply medical device fully around intrauterine surgery area
  Arms: Adept

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Mediclore®, as an antiadhesive barrier, which is made of Poloxamer, Gelatin and Chitosan.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Gynecological disease (benign disease)
* Patients who Written informed consent
* Patients without clinically significant lab

Exclusion Criteria:

* having enrolled another clinical trials within 1 month
* Immunosuppression or autoimmune disease
* Anticoagulant, general steroids within a week from surgery
* Serious diseases (heart failure, renal failure, liver failure, uncontrolled hypertension, diabetes mellitus, coagulation deficiencies)
* Patients with previous history of surgery at the same operate site

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-07 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
adhesion rate | 4 weeks after surgery
  4 weeks after surgery, finding adhesion using visceral slide test

SECONDARY OUTCOMES:
Incidence of adhesion symptoms | 4 weeks after surgery
  4 weeks after surgery, Identifying adhesion sysmptoms using Questionnaire
adverse event | 4 weeks after surgery
  identifying adverse events after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Seoutl National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided